CLINICAL TRIAL: NCT01484574
Title: A Non-randomized, Open Label, Multicentric, Dose Ranging , Phase II Study Assessing the Efficacy and Safety of Intramuscular Administration of Stempeucel - CLI™ (ex Vivo Cultured Adult Bone Marrow Derived Allogeneic Mesenchymal Stem Cells) in Patients With Critical Limb Ischemia Due to Buerger's Disease
Brief Title: A Clinical Trial to Study the Efficacy and Safety of Different Doses of Bone Marrow Derived Mesenchymal Stem Cells in Patients With Critical Limb Ischemia Due to Buergers Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stempeutics Research Pvt Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SRPL/CLI/10-11/001
Record Dates: First submitted 2011-11-27; First posted 2011-12-02 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Critical Limb Ischemia; Buerger's Disease
Keywords: Critical limb ischemia; Buerger's disease; Critical limb ischemia due to Buerger's disease
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Thromboangiitis Obliterans

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low dose (Experimental): Stempeucel - CLI will be administered at the lowest dose
  Interventions: Biological: Allogeneic Mesenchymal Stem Cells
- Intermediate dose (Experimental): Stempeucel - CLI will be administered at intermediate dose
  Interventions: Biological: Allogeneic Mesenchymal Stem Cells
- Control arm (No Intervention): Standard protocol of care alone

INTERVENTIONS:
Biological: Allogeneic Mesenchymal Stem Cells — Single intramuscular administration of low dose of stem cells
  Other Names: Stempeucel - CLI
  Arms: Low dose
Biological: Allogeneic Mesenchymal Stem Cells — Single intramuscular administration of intermediate dose of stem cells
  Other Names: Stempeucel - CLI
  Arms: Intermediate dose

SUMMARY:
This is an open label, non-randomized, dose ranging study to evaluate the safety and efficacy of different doses of Stempeucel in critical limb ischemia patients.

ELIGIBILITY:
Inclusion Criteria:

* Buerger's disease as diagnosed by Shionoya criteria
* Males or females (willing to use accepted methods of contraception during the course of the study) in the age group of 18-65 yrs
* Established CLI in the study limb, clinically and hemodynamically confirmed as per Rutherford- III-5
* Patients in Rutherford- III-6 if gangrene extending maximally up to the head of metatarsal but limited to toes (Patients with wet gangrene must undergo wound debridement / amputation before screening)
* Patients having infrapopliteal occlusive disease with rest pain and ischemic ulcer/necrosis, who are not eligible for or have failed traditional revascularization treatment as per the investigators judgment (No option patients)
* Ankle Brachial Pressure Index (ABPI) ≤ 0.6 or ankle pressure ≤ 50 mm Hg or TcPO2 ≤ 40 mmHg in the foot of the study limb
* Patients who are able to understand the requirements of the study, and willing to provide voluntary written informed consent and video consent, abide by the study requirements, and agree to return for required follow-up visits

Exclusion Criteria:

* Patients with CLI indicated for major amputation during screening
* Atherosclerotic PAD
* Ulcers with exposure of tendon and/bone in the shin region
* Previous above transmetatarsal amputation in study limb
* Any Lumbar sympathectomy procedure performed less than 90 days prior to the screening
* Patients with gait disturbance for reasons other than CLI
* Diagnosis of diabetes mellitus (type 1 or type 2)
* Patients having left ventricular ejection fraction < 35%
* Patients suffering from clinically relevant peripheral neuropathy
* History of Stroke or myocardial infarction
* Patients who are contraindicated for MRA
* Patients with deep vein thrombosis in any limb
* Patients who have clinically serious and/or unstable inter-current infection, medical illnesses or conditions that are uncontrolled or whose control, in the opinion of the Investigator, may be jeopardized by participation in this study or by the complications of this therapy
* Documented terminal illness or cancer or any concomitant disease process with a life expectancy of <1 year
* Patients already enrolled in another investigational drug trial or completed within 3 months or those who have participated in any stem cell clinical trial
* Patient with known hypersensitivity to the constituents of the IMP - dimethyl sulfoxide (DMSO) or human serum albumin (HSA)
* History of severe alcohol or drug abuse within 3 months of screening
* Hb% < 10 gm% for males, Hb% < 9 gm% for females, serum creatinine ≥ 2mg%, serum Total Bilirubin ≥2mg%
* Pregnant and lactating women
* Patients tested positive for HIV 1, HCV, HBV, CMV, RPR

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2012-01; Primary Completion 2014-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Relief of the rest pain | 6 months
  Rest pain will be measured using rest pain scale (0 to10)
Healing of ulcerations or reduction of ulcer area in the target limb | 6 months
  Complete ulcer healing defined as complete epithelisation of ulcer and partial ulcer healing as at least 30% decrease in ulcer size.
Relief of the rest pain | 24 months
  Rest pain will be measured using rest pain scale (0 to 10)
Healing of ulcerations or reduction of ulcer area in the target limb | 24 months
  Complete ulcer healing defined as complete epithelisation of ulcer and partial ulcer healing as at least 30% decrease in ulcer size.

SECONDARY OUTCOMES:
Pain free walking distance | 6 and 24 months
Major amputation free survival | 6 and 24 months
Ankle brachial pressure index (ABPI) - measured by Doppler | 6 and 24 months
Increase in transcutaneous partial oxygen pressure (TcPO2) | 6 and 24 months
Quality of life by King's College VascuQOL questionnaire | 6 and 24 months
Angiogenesis - collateral blood vessels by Magnetic resonance angiogram (MRA) | 6 and 24 months
The type of adverse events AE(s), number of AE(s) and proportion of patients with AE(s). | 6 and 24 months
Assessment of clinical laboratory parameters | 6 and 24 months
Physical examination findings and assessment of vital signs | 6 and 24 months
Assessment of electrocardiogram (ECG) parameters | 6 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr Anirban Chatterjee, Principal Investigator — AMRI Hospital; Dr Anita Dhar, Principal Investigator — All India Institute of Medical Sciences; Dr Rajkumar M, Principal Investigator — Stanley Medical College; Dr Radhakrishnan R, Principal Investigator — Sri Ramchandra Medical College; Dr Vidyasagaran T, Principal Investigator — Madras Medical College; Dr Alfred Augustine, Principal Investigator — KMC, Mangalore; Dr Sanjay Desai, Principal Investigator — M. S. Ramaiah Medical College; Dr Rajiv Parakh, Principal Investigator — Medanta - The Medicity; Dr Santanu Dutta, Principal Investigator — Nightingale Hospital; Dr Murali Krishna, Principal Investigator — Sri Jayadeva Institute of Cardiovascular Sciences & Research
Locations (10):
- India (10):
  - Division of Peripheral Vascular and Endovascular Sciences, Medanta - The Medicity, Gurgaon, Haryana
  - Department of Vascular and Endovascular Surgery, M. S. Ramaiah Medical College and Hospitals, Bangalore, Karnataka
  - Peripheral Vascular Surgery, Sri Jayadeva Institute of Cardiovascular Sciences & Research, Bangalore, Karnataka
  - Department of Surgery, KMC, Mangalore, Mangalore, Karnataka
  - Department of Surgical Disciplines, All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi
  - Department of Vascular Surgery, Madras Medical College, Chennai, Tamil Nadu
  - Department of Vascular Surgery, Sri Ramchandra Medical College, Chennai, Tamil Nadu
  - Department of Vascular Surgery, Stanley Medical College, Chennai, Tamil Nadu
  - Department of Vascular Surgery, AMRI Hospital, Kolkata, West Bengal
  - Nightingale Hospital, Kolkata, West Bengal